CLINICAL TRIAL: NCT04994678
Title: EFFECT OF VIRTUAL REALITY-BASED EXERCISE REGIME ON POSTURAL STABILITY AND GAIT DYNAMICS
Brief Title: EFFECT OF VIRTUAL REALITY BASED EXERCISE REGIME ON POSTURAL STABILITY AND GAIT DYNAMICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2021/1
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Fall

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to interventional group (virtual Reality Training Group) and Control Group (Aerobic Training Group) for whole duration of study.
Who Masked: Outcomes Assessor
Masking Description: Single blinded study with random allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Training Group (Experimental): VR training system will be setup in multidisciplinary lab of Foundation University Institute of Rehabilitation Sciences Foundation University Islamabad. Display will be provided on 55 inch LED TV with audio feedback. Display will be at height of 5 feet from floor and at distance of 6 feet from Subject. The Virtual reality based training group will receive a game based virtual reality training via XBOX 360 or wii fit balance games. Particiapants will be required to physically move to move avatar on screen to rapidly leaning away, squat to avoid overhead obstacles and try small jump to avoid lower obstacles, single leg stance, in addition person will required to do half squatting, side to side jumps and vertical jumps. Treatment will be provided 3 times a week for 6 weeks with each session lasting for 30-50 minutes. Progressively challenge will be increased.
  Interventions: Other: Virtual Reality Training
- Moderate Aerobic Exercise Training Group (Active Comparator): Moderate aerobic exercise training will be provided using motorized tread mill and stationary/recombinent cycle. Treatment will be provided for 30-50 minutes 3 times a week for 6 weeks.
  Interventions: Other: Moderate Aerobic Exercise Training

INTERVENTIONS:
Other: Virtual Reality Training — The Virtual reality based training group will receive a game based virtual reality training via XBOX 360or wii fit balance games. Player will be required to rapidly leaning away, squat to avoid overhead obstacles and try small jump to avoid lower obstacles, single leg stance, in addition person will required to do half squatting, side to side jumps and vertical jumps. Treatment will be provided 3 times a week or 6 weeks with each session lasting for 30-50 minutes. Progressively challenge will be increased.
  Arms: Virtual Reality Training Group
Other: Moderate Aerobic Exercise Training — Moderate intensity continuous Aerobic exercises (Recombinant/Stationary cycling for 10-15 min with progression followed by treadmill walking for 10-15 min with progression, as well as stepping and Jogging). The session will be preceded by 5-7 minute warm-up & 7-10 min cool-down.
  Arms: Moderate Aerobic Exercise Training Group

SUMMARY:
People worldwide are living longer. Today, for the first time in history, most people can expect to live into their sixties and beyond. By 2050, the world's population aged 60 years and older is expected to total 2 billion, up from 900 million in 2015. Today, 125 million people are aged 80 years or older. By 2050, there will be almost this many (120 million) living in China alone, and 434 million people in this age group worldwide. By 2050, 80% of all older people will live in low- and middle-income countries.

As we age, we lose balance function through loss of sensory elements, the ability to integrate information and issue motor commands, and because we lose musculoskeletal function. Diseases common in aging populations lead to further deterioration in balance function in some patients.

study aims to determine the Effect of Virtual Reality exercise regimen on postural stability and gait dynamics in elderly population. By obtaining these results we can recommend and effective balance training regime which can be implemented in health care system and hence resulting in decrease fall events in geriatric population and also reduce fall related health care financial burden on economy.

DETAILED DESCRIPTION:
Elderly population presenting in Emergency Room are responsible for increased consumption of health care resources but they are easily identifiable population who have high risk of fall. Older people have the highest risk of death or serious injury arising from a fall and the risk increases with age. For example, in the United States of America, 20-30% of older people who fall suffer moderate to severe injuries such as bruises, hip fractures, or head trauma. This risk level may be in part due to physical, sensory, and cognitive changes associated with ageing, in combination with environments that are not adapted for an ageing population.

Falls and falls risks can be reduced through systematic risk identification and targeted intervention, including a combination of clinical and community-based interventions. Multiple evidence-based community programs have been shown to reduce falls and/or falls risk factors.

Using the gaming with the biofeedback system, such as the virtual reality (VR) system, is widely used for rehabilitation. It is due to the fact that the VR system can make the treatment more interesting, reduce the difficulty of rehabilitation, and increase safety In this study participants will be divided in 2 groups.

1 group will recieve Virtual reality Training and other group will Recieve Aerobic Training.

Treatment will be given 3 times a week for 6 weeks by researcher with each session lasting 30-50 Minutes.

Assessment of postural stability and other outcome measures will be done after every two weeks till Terminal assessment after 6 weeks of treatment by same Physical Therapist who did initial Assessment. In addition, assessment gait parameters will be done at baseline and at end of trial.

ELIGIBILITY:
Inclusion Criteria

* Elderly Population the age of 55 Years
* Either Gender
* Not performing any Systematic strength or Aerobic Training Exclusion Criteria
* Severe orthopedic, cardiovascular pulmonary disease.
* History of Surgery & Severe Trauma of Lower extremity.
* Other musculoskeletal Disorders (Scoliosis & Lordosis)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Postural Stability Assessment | 6 weeks
  Postural stability assessment will be done via use of Biodex balance system SD.
Gait Parameters | 6 weeks
  Spatial and temporal Gait Parameters including step width, step length, stride length, cadence.

SECONDARY OUTCOMES:
Mobility | 6 weeks
  Mobility will be assessed using time up and go test
Functional Lower Extremity Strength | 6 weeks
  Functional Lower Extremity Strength will be assessed using 5 times sit to stand
Aerobic capacity | 6 weeks
  Aerobic capacity will be assessed using 6minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ehab Azim, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No